CLINICAL TRIAL: NCT01455077
Title: Validation of a Portable Monitoring System for the Diagnosis of Obstructive Sleep Apnea Syndrome in Patients With Level II and III Obesity
Brief Title: Portable Monitoring Device for the Diagnosis of Sleep Apnea in Obese Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Associacao Fundo de Incentivo a Psicofarmcologia (Other)
Collaborators: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Prof. Dr. Lia Azeredo-Bittencourt, MD, PhD, associate professor, Associacao Fundo de Incentivo a Psicofarmcologia
Other Study IDs: CEP0290/11; Portable monitoring system for; STD obesity
Record Dates: First submitted 2011-10-15; First posted 2011-10-19 (Estimated); Last update posted 2011-10-19 (Estimated); Status verified 2011-10

CONDITIONS: Obstructive Sleep Apnea Syndrome; Obesity
Keywords: obesity; sleep apnea; portable monitoring
MeSH Terms: conditions — Sleep Apnea, Obstructive; Obesity; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Obese patients: BMI > 35

SUMMARY:
Introduction The portable monitoring system (PMS) recording of cardiopulmonary parameters (level III of ASDA) has been validated in subjects with high probability of Obstructive Sleep Apnea (OSA) without comorbidities.

However, there is not any study evaluating this system when OSA is associated with morbid obesity, so the validation of PMS will be very useful in order to properly work-up this highly risk population.

Objective:

To evaluate the accuracy of level III type of PMS - Stardust™" (STD), on patients with level II and III of obesity and high clinical suspicion of OSA.

Methods:Participants with BMI > 35 kg/m2 and with suspicion of OSA will consecutively be selected from an Outpatients Sleep Clinic of UNIFESP. They will be randomized for the following order of recordings:

1) STD at home for 1 night 2) STD in the sleep lab simultaneous to PSG. AHI will be taken for subsequent analysis:a) AHI PSG b) AHI STD -lab and c) AHI STD- home.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 35
* Complaints of snoring, sleep apnea, daytime sleepiness

Exclusion Criteria:

* use of home oxygen
* other sleep diseases
* inability to perform PSG

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults BMI > 35 Male and female
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-07 (Actual); Study Completion 2012-01 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Associacao Fundo de Incentivo a Psicofarmacologia, São Paulo, São Paulo, Brazil